CLINICAL TRIAL: NCT03055676
Title: A Randomized Prospective Multicenter Trial of Early Versus Late Drain Removal After Pancreaticoduodenectomy
Brief Title: Prospective Multicenter Trial of Early Versus Late Drain Removal After Pancreaticoduodenectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Peking University First Hospital (Other); Chinese PLA General Hospital (Other); Xuanwu Hospital, Beijing (Other); Beijing Chao Yang Hospital (Other); Beijing Tongren Hospital (Other); Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PUMCH-GS05
Record Dates: First submitted 2017-02-14; First posted 2017-02-16 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Pancreaticoduodenectomy; Drainage
Keywords: Pancreaticoduodenectomy; Time of drain removal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Early drain removal (Experimental): Removing drain(s) on postoperative day 3 (n = 166)
  Interventions: Other: Early drain removal
- Late drain removal (Active Comparator): Removing drain(s) on postoperative day 5 or later (n = 166)
  Interventions: Other: Late drain removal

INTERVENTIONS:
Other: Early drain removal — Removing drain(s) on postoperative day 3
  Arms: Early drain removal
Other: Late drain removal — Removing drain(s) on postoperative day 5 or later
  Arms: Late drain removal

SUMMARY:
The aim of this randomized prospective multicenter study is to demonstrate the hypothesis that early removal of drain could reduce the incidence of major complications (grade 2-4) after pancreaticoduodenectomy (PD) , when compared with later removal of drain.

DETAILED DESCRIPTION:
The objective of this randomized prospective multicenter study is to investigate the association between the time of removal of drain after pancreaticoduodenectomy (PD) and incidence of major complications (grade 2-4 complications). The investigators unite six pancreatic surgery center in Beijing. Patients who underwent pancreaticoduodenectomy (PD) or pylorus-preserving pancreaticoduodenectomy (PPPD) with low to moderate risk of post-operative pancreatic fistula (POPF) are recruited into the study. After obtaining informed consent, eligible patients are randomly allocated to early or late drain removal group on POD 3. In the group A, drain(s) are removed on POD 3, whereas in group B drain is removed on POD 5 or beyond. The primary outcomes are the incidence of sum of grade 2-4 complications, the secondary outcomes include grade B/C POPF, intra-abdominal infeciton, delayed gastric emptying, post-operative bleeding, in-hospital stay, total medical cost and comprehensive complication index (CCI).

ELIGIBILITY:
Inclusion Criteria:

1. PD with or without pylorus preserving;
2. Age between 18 and 75 years;
3. Drain amylase on POD 1 and 3 less than 5000 U/L;
4. Drain output within POD 3 less than 300 ml per day.

Exclusion Criteria:

1. Vascular reconstruction using an artificial graft;
2. Grade B/ C postoperative bleeding, evident anastomosis leakage within 3 days after surgery;
3. Refusale to participate in after signed informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 319 (Actual)
Dates: Start 2017-01; Primary Completion 2020-03 (Actual); Study Completion 2020-04 (Actual)

PRIMARY OUTCOMES:
The sum of grade 2- 4 complications | Up to postoperative 90 days
  The severity of complication was measured by Clavein Dindo classifications and grade 2- 4 complications always affect the recovery of the patients significantly.However, the death case (grade 5 complication) is rare now for PD in high volume centers. According to our single center study, early drain removal could reduce the rate of grade 2-4 complications by 12% for the patients undergoing major pancreatectomy.

SECONDARY OUTCOMES:
Intra-abdominal bleeding | Up to postoperative 90 days
  The International Study Group of Pancreatic Surgery (ISGPS) definition: Blood loss through abdominal drains or nasogastric tube;hematemesis or melena; clinical deterioration of the patient; unexplained hypotension or tachycardia; or laboratory findings such as a decreasing hemoglobin concentration.
Delayed gastric emptying | Up to postoperative 90 days
  The International Study Group of Pancreatic Surgery (ISGPS) definition: Inability to return to a standard diet by the end of the first postoperative week with prolonged nasogastric intubation.
Grade B/C complications | Up to postoperative 90 days
  The International Study Group of Pancreatic Surgery (ISGPS) definition
Length of hospital stay (day) | Up to postoperative 90 days
  Participants will be followed for the duration of hospital stay, an expected average of 2 weeks.
Comprehensive complication index (CCI) | Up to postoperative 90 days
  integrates all complications of the Clavien-Dindo classification (CDC) and offers a metric approach to measure morbidity.
Interventional treatment | Up to postoperative 90 days
  interventional treatment for any complication.
Total medical expenses | Up to postoperative 90 days
  Total medical expenses during hospitalization.
Any other single intem of grade 2-4 complication | Up to postoperative 90 days
  Clavein Dindo Classification is adopted.

CONTACTS AND LOCATIONS:
Overall Officials: Menghua Dai, M.D., Study Chair — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
After this multicenter randomized clinical trail complete, the results of this study will be submitted to and published in a peer-reviewing journal. Other researchers can assess our article through electronic database, such as Medline/PubMed.

REFERENCES:
- [Background] Van Buren G 2nd, Bloomston M, Hughes SJ, Winter J, Behrman SW, Zyromski NJ, Vollmer C, Velanovich V, Riall T, Muscarella P, Trevino J, Nakeeb A, Schmidt CM, Behrns K, Ellison EC, Barakat O, Perry KA, Drebin J, House M, Abdel-Misih S, Silberfein EJ, Goldin S, Brown K, Mohammed S, Hodges SE, McElhany A, Issazadeh M, Jo E, Mo Q, Fisher WE. A randomized prospective multicenter trial of pancreaticoduodenectomy with and without routine intraperitoneal drainage. Ann Surg. 2014 Apr;259(4):605-12. doi: 10.1097/SLA.0000000000000460. PMID 24374513
- [Background] Kawai M, Tani M, Terasawa H, Ina S, Hirono S, Nishioka R, Miyazawa M, Uchiyama K, Yamaue H. Early removal of prophylactic drains reduces the risk of intra-abdominal infections in patients with pancreatic head resection: prospective study for 104 consecutive patients. Ann Surg. 2006 Jul;244(1):1-7. doi: 10.1097/01.sla.0000218077.14035.a6. PMID 16794381
- [Background] Bassi C, Molinari E, Malleo G, Crippa S, Butturini G, Salvia R, Talamini G, Pederzoli P. Early versus late drain removal after standard pancreatic resections: results of a prospective randomized trial. Ann Surg. 2010 Aug;252(2):207-14. doi: 10.1097/SLA.0b013e3181e61e88. PMID 20622661
- [Background] Wente MN, Bassi C, Dervenis C, Fingerhut A, Gouma DJ, Izbicki JR, Neoptolemos JP, Padbury RT, Sarr MG, Traverso LW, Yeo CJ, Buchler MW. Delayed gastric emptying (DGE) after pancreatic surgery: a suggested definition by the International Study Group of Pancreatic Surgery (ISGPS). Surgery. 2007 Nov;142(5):761-8. doi: 10.1016/j.surg.2007.05.005. PMID 17981197
- [Background] Bassi C, Dervenis C, Butturini G, Fingerhut A, Yeo C, Izbicki J, Neoptolemos J, Sarr M, Traverso W, Buchler M; International Study Group on Pancreatic Fistula Definition. Postoperative pancreatic fistula: an international study group (ISGPF) definition. Surgery. 2005 Jul;138(1):8-13. doi: 10.1016/j.surg.2005.05.001. PMID 16003309
- [Background] Wente MN, Veit JA, Bassi C, Dervenis C, Fingerhut A, Gouma DJ, Izbicki JR, Neoptolemos JP, Padbury RT, Sarr MG, Yeo CJ, Buchler MW. Postpancreatectomy hemorrhage (PPH): an International Study Group of Pancreatic Surgery (ISGPS) definition. Surgery. 2007 Jul;142(1):20-5. doi: 10.1016/j.surg.2007.02.001. PMID 17629996
- [Derived] Dai M, Liu Q, Xing C, Tian X, Cao F, Tang W, Lv S, Ma Y, Zhang D, Kleeff J, Yang Y, Liu R, He Q, Li F, Li G, Guo J, Liao Q, Zhao Y. Early Drain Removal is Safe in Patients With Low or Intermediate Risk of Pancreatic Fistula After Pancreaticoduodenectomy: A Multicenter, Randomized Controlled Trial. Ann Surg. 2022 Feb 1;275(2):e307-e314. doi: 10.1097/SLA.0000000000004992. PMID 34117153